CLINICAL TRIAL: NCT01507805
Title: Effects of Electroacupuncture Preconditioning on Outcomes of the Geriatric Patients With Coronary Heart Disease Undergoing Non-cardiac Surgery
Brief Title: Electroacupuncture Preconditioning on Geriatric Noncardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: csyxijing
Record Dates: First submitted 2011-12-13; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-02

CONDITIONS: Coronary Heart Disease
Keywords: Electroacupuncture; preconditioning; Non-cardiac surgery; Coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EA preconditioning (Experimental): electroacupuncture five days pre-operation
  Interventions: Device: EA preconditioning
- Sham EA preconditioning (Sham Comparator): Patients treated with sham EA preconditioning Intervention
  Interventions: Device: sham EA preconditioning

INTERVENTIONS:
Device: EA preconditioning — EA preconditioning group was treated at bilateral Neiguan(PC 6)，Lieque(LU 7)and Yunmen(LU 2)with electrical stimulation(5-30 Hz，2．34-6．24 mA，30 min)for 5 consecutive days before surgery
  Other Names: Huantuo sdz-Ⅱ,Suzhou Medical Limit
  Arms: EA preconditioning
Device: sham EA preconditioning — Patients in Sham EA preconditioning group was treated at bilateral Neiguan(PC 6)，Lieque(LU 7)and Yunmen(LU 2)without electrical stimulation(5-30 Hz，2．34-6．24 mA，30 min)for 5 consecutive days before surgery
  Arms: Sham EA preconditioning

SUMMARY:
The purpose of this study is to observe whether the electroacupuncture (EA) preconditioning for five days before operation can improve the outcomes of patients with coronary heart disease undergoing geriatric non-cardiac surgery.

DETAILED DESCRIPTION:
BACKGROUND:

With the development of surgical techniques, more and more people with coronary heart disease underwent non-cardiac surgery, which include abdominal, urologic, orthopedic surgeries. Due to the vulnerable heart function, geriatric patients suffer high incidence of cardiovascular events during the peri-operative period. Some studies found that EA preconditioning have a protective effect for the patients underwent Cardiac surgery. But non one addresses the effects of EA preconditioning on the outcomes of the patients with coronary heart disease who undergo non-cardiac surgery.

DESIGNING:

The patients with coronary heart disease who will receive abdominal surgery will be randomly assigned into EA preconditioning group and control group. The patients in EA preconditioning group was treated at bilateral Neiguan (PC 6)，Lieque (LU 7) and Yunmen (LU 2) with electrical stimulation (5-30 Hz，2．34-6．24 mA，30 min) for 5 consecutive days before surgery．Before operation and before surgery, after surgery, 24h, 72h post surgery, all patients will be subjected to test the serum level of c-reactive protein and Troponin I. The EEG and heart ultrasonic exam will be used to evaluate the condition and function of heart before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective abdominal surgery with coronary heart disease

Exclusion Criteria:

* serious bradycardiac arrythmia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-06 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The change of myocardial ischemic injury markers,including serum level of c-reactive protein and Troponin I | 10 minutes before EA, 10 minutes pre-operation,the day of post-operation, 24hours post-operation, 72 hours post-operation
  to observe the change of the level of multiple myocardial ischemic injury markers at the different time points.

SECONDARY OUTCOMES:
The change of ST segment of EEG at different time points | 10 minutes before EA, 10 minutes pre-operation,the day of post-operation, 24hours post-operation, 72 hours post-operation
Cardiac ultrasonic scan | five days pre-operation , five days post-operation
  be aware of cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyang Chen, M.D., Principal Investigator — Xijing Hospital, the Fourth Military Medical University
Locations (1):
- Xijing hospital, Xi'an, Shannxi, China